CLINICAL TRIAL: NCT00849017
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of Two Dose Levels of Albiglutide Compared With Placebo in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy Study of Albiglutide in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112756
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: placebo; albiglutide; monotherapy; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- albiglutide (Experimental): albiglutide weekly injection
  Interventions: Biological: albiglutide
- placebo (Placebo Comparator): albiglutide matching placebo
  Interventions: Biological: placebo
- albiglutide up-titration (Experimental): albiglutide weekly injection uptitration at week 12
  Interventions: Biological: albiglutide uptitration

INTERVENTIONS:
Biological: albiglutide — albiglutide weekly injection
  Arms: albiglutide
Biological: albiglutide uptitration — albiglutide uptitration at week 12
  Arms: albiglutide up-titration
Biological: placebo — matching albiglutide placebo weekly injection
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether albiglutide is effective in the treament of patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI 20-45kg/m2 inclusive

Exclusion Criteria:

* females who are pregnant, lactating, or <6 weeks post-partum
* CHF NYHA class III-IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (221):
- United States (208):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bull Shoals, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Indio, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Middletown, Delaware
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Crescent Springs, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Interlochen, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Broken Bow, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Hainesport, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Chadbourn, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Thornville, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Melrose Park, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Crossville, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Virgina Beach, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Richland, Washington
  - GSK Investigational Site, Selah, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Mexico (12):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Puebla City, Puebla
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Cuernavaca
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Nezahualcóyotl
  - GSK Investigational Site, Torreón
- GSK Investigational Site, Parow, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Home PD, Ahren B, Reusch JEB, Rendell M, Weissman PN, Cirkel DT, Miller D, Ambery P, Carr MC, Nauck MA. Three-year data from 5 HARMONY phase 3 clinical trials of albiglutide in type 2 diabetes mellitus: Long-term efficacy with or without rescue therapy. Diabetes Res Clin Pract. 2017 Sep;131:49-60. doi: 10.1016/j.diabres.2017.06.013. Epub 2017 Jun 15. PMID 28683300
- [Derived] Nauck MA, Stewart MW, Perkins C, Jones-Leone A, Yang F, Perry C, Reinhardt RR, Rendell M. Efficacy and safety of once-weekly GLP-1 receptor agonist albiglutide (HARMONY 2): 52 week primary endpoint results from a randomised, placebo-controlled trial in patients with type 2 diabetes mellitus inadequately controlled with diet and exercise. Diabetologia. 2016 Feb;59(2):266-74. doi: 10.1007/s00125-015-3795-1. Epub 2015 Nov 17. PMID 26577795
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Young MA, Wald JA, Matthews JE, Yang F, Reinhardt RR. Effect of renal impairment on the pharmacokinetics, efficacy, and safety of albiglutide. Postgrad Med. 2014 May;126(3):35-46. doi: 10.3810/pgm.2014.05.2754. PMID 24918790
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 4 week Run-in/Stabilization Period were then randomized to a 156-week Treatment Period, followed by 8 weeks of post-treatment follow-up. A total of 479 par. were screened; 309 par. were randomized, and 301 par. received >=1 treatment dose.
Groups:
- Placebo: Participants received matching placebo as a subcutaneous injection weekly via a fully disposable pen injector system. Participants did not receive investigational product during the Follow-up Period.
- Albiglutide 30 mg: Participants received albiglutide 30 milligrams (mg) as a subcutaneous injection weekly via a fully disposable pen injector system. Participants did not receive investigational product during the Follow-up Period.
- Albiglutide 50 mg: Participants received albiglutide 30 mg from Baseline to Week 12 with a forced blinded uptitration to 50 mg at Week 12 as a subcutaneous injection weekly via a fully disposable pen injector system. Participants did not receive investigational product during the Follow-up Period.
Period: Treatment Period (156 Weeks)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Started | 101 | 101 | 99
Completed | 58 | 68 | 57
Not Completed | 43 | 33 | 42
Not completed — Adverse Event | 5 | 6 | 15
Not completed — Noncompliance | 3 | 3 | 4
Not completed — Lost to Follow-up | 10 | 7 | 8
Not completed — Withdrawal by Subject | 18 | 14 | 11
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Termination of Study/ Site by GSK | 3 | 1 | 1
Not completed — Increased Calcitonin | 1 | 0 | 0
Not completed — Physician Discontinued-Thrombocytopenia | 1 | 0 | 0
Not completed — Participant Moved to Africa | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Participant Decided to Move Out of State | 0 | 0 | 1
Period: Follow-up Period (8 Weeks)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Started | 101 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 101 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 99 (Participants withdrawing from the Treatment Period entered the Follow-up Period.)
Completed | 76 | 83 | 74
Not Completed | 25 | 18 | 25
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Noncompliance | 2 | 1 | 0
Not completed — Lost to Follow-up | 13 | 12 | 16
Not completed — Did Not Enter Follow-up Period | 1 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Termination of Study/ Site by GSK | 3 | 1 | 1
Not completed — Participant Relocating to Africa | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg | Total
Number analyzed (Participants) | 101 | 101 | 99 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.68) | 53.6 (10.89) | 52.0 (11.75) | 52.9 (11.43)
Gender [Count of Participants; unit: Participants]
  Female | 43 | 43 | 49 | 135
  Male | 58 | 58 | 50 | 166
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 14 | 10 | 14 | 38
  American Indian or Alaskan Native | 3 | 1 | 1 | 5
  Asian - Central/South Asian Heritage | 0 | 1 | 1 | 2
  Asian - East Asian Heritage | 2 | 0 | 0 | 2
  Asian - Japanese Heritage | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 2 | 6
  White - Arabic/North African Heritage | 0 | 2 | 3 | 5
  White - White/Caucasian/European Heritage | 77 | 85 | 78 | 240

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: Glycated hemoglobin (HbA1c) is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 52 minus the value at BL. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, history of prior myocardial infarction (yes versus no), and age category (<65 years versus ≥65 years) as factors and Baseline HbA1c as a continuous covariate. The last observation carried forward (LOCF) method was used to impute missing post-BL HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 98 | 100 | 97
Percentage of HbA1c in the blood | 0.15 (0.097) | -0.70 (0.096) | -0.89 (0.097)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 30 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.11 to -0.58]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 50 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.04, 95% CI 2-sided [-1.31 to -0.77]

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 104 and 156
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Weeks 104 and 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 99 | 100 | 97
Percentage of HbA1c in the blood
  Week 104, n=21, 39, 42 | -0.40 (0.676) | -0.93 (1.027) | -1.18 (0.909)
  Week 156, n=14, 30, 32 | -0.61 (0.644) | -0.96 (0.968) | -1.07 (0.887)

3. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: FPG >=280 milligrams/deciliter (mg/dL) between >=Week 2 and <Week 4; FPG >=250 mg/dL between >=Week 4 and <Week 12; HbA1c >=8.5% and a <=0.5% reduction from Baseline between >=Week 12 and <Week 24; HbA1c >=8.5% between >=Week 24 and <Week 48; HbA1c >=8.0% between >= Week 48 and <Week 156. Participants could have been rescued at any time on or after Week 2. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus 1 day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus 1 day for participants not requiring rescue. This time was divided by 7 to express the result in weeks.
Time Frame: From the start of study medication until the end of the treatment (up to Week 156)
Population: IIT Population. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 99 | 100 | 97
Weeks | 49.71 [32.14 to 67.29] | 118.43 [79.43 to NA] — The 95% CI upper bound is not a available because it is beyond study duration. | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline weight + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 99 | 100 | 97
Millimoles per liter (mmol/L) | 1.00 (0.239) | -0.88 (0.237) | -1.38 (0.241)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 156
Description: The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline FPG minus the Baseline FPG.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 14 | 29 | 32
Millimoles per liter (mmol/L) | -0.23 (0.794) | -1.31 (1.761) | -1.83 (2.012)

6. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 52
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 52) were assessed.
Time Frame: Week 52
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 98 | 100 | 97
Participants
  Week 52, HbA1c <6.5% | 10 | 25 | 24
  Week 52, HbA1c <7.0% | 21 | 49 | 39
  Week 52, HbA1c <7.5% | 34 | 59 | 62

7. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 156
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 156) were assessed.
Time Frame: Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed. This analysis used observed HbA1c values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 14 | 30 | 32
Participants
  Week 156, HbA1c <6.5% | 6 | 10 | 11
  Week 156, HbA1c <7.0% | 8 | 18 | 19
  Week 156, HbA1c <7.5% | 13 | 24 | 29

8. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with prerescue values. Based on ANCOVA: change = treatment + Baseline weight + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 99 | 100 | 97
Kilograms | -0.66 (0.428) | -0.39 (0.424) | -0.86 (0.432)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 156
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants who were available at the indicated time points were analyzed. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 14 | 30 | 31
Kilograms | -2.91 (5.213) | -1.32 (5.123) | -2.24 (5.589)

10. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose Profile Parameter-4 Hour C-peptide AUC
Description: Changes from Baseline at Week 52 in postprandial parameters after a mixed-meal (MM) tolerance test were analyzed. Post prandial blood glucose parameter analyzed was 4 hour c-peptide AUC. The AUC was determined using the trapezoidal method using measurements until 4 hours following the meal. The standardized AUC is the total AUC divided by elapsed time. Those parameters were analyzed analogous to the primary endpoint using an ANCOVA model with treatment group as a factor, and corresponding Baseline postprandial profile as a continuous covariate. This analysis used observed values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 52
Population: MM Population: all participants who participated in the MM tolerance test substudy and who had valid Baseline assessments and Week 52 assessments for at least 1 of the MM lab parameter of C-peptide.
Measure: Least Squares Mean (Standard Error); unit: Nanomoles/Liter (nmol/L)
Groups:
- Albiglutide 30 mg Weekly: Participants received albiglutide 30 milligrams (mg) as a subcutaneous injection weekly via a fully disposable pen injector system. Participants did not receive investigational product during the Follow-up Period.
- Albiglutide 50 mg Weekly: Participants received albiglutide 30 mg from Baseline to Week 12 with a forced blinded uptitration to 50 mg at Week 12 as a subcutaneous injection weekly via a fully disposable pen injector system. Participants did not receive investigational product during the Follow-up Period.
Arm/Group | Placebo | Albiglutide 30 mg Weekly | Albiglutide 50 mg Weekly
Number analyzed (Participants) | 8 | 16 | 20
Nanomoles/Liter (nmol/L) | 0.05 (0.165) | 0.03 (0.122) | 0.08 (0.108)

11. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose Profile Parameter- 4 Hour Blood Glucose AUC
Description: Changes from Baseline at Week 52 in postprandial parameters after a mixed-meal (MM) tolerance test were analyzed. Post prandial blood glucose parameter analyzed was: 4 hour blood glucose area under urve AUC The AUC was determined using the trapezoidal method using measurements until 4 hours following the meal. The standardized AUC is the total AUC divided by elapsed time. Those parameters were analyzed analogous to the primary endpoint using an ANCOVA model with treatment group as a factor, and corresponding Baseline postprandial profile as a continuous covariate. This analysis used observed values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 52
Population: MM Population: all participants who participated in the MM tolerance test substudy and who had valid baseline assessments and Week 52 assessments for at least 1 of the MM lab parameter of glucose. The MM tolerance test was performed only in those participants who additionally consented to participate in.
Measure: Least Squares Mean (Standard Error); unit: Nanomoles/Liter (nmol/L)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 8 | 18 | 19
Nanomoles/Liter (nmol/L) | -0.51 (0.630) | -1.74 (0.414) | -2.05 (0.407)

12. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose Profile Parameters-4 Hour Insulin AUC and 4 Hour Proinsulin AUC
Description: Changes from Baseline at Week 52 in postprandial parameters after a mixed-meal (MM) tolerance test were analyzed. Post prandial blood glucose parameters analyzed were: 4-hour insulin AUC (4 hr Ins AUC), and 4-hour proinsulin AUC (4 hr pro-Ins AUC). The AUC was determined using the trapezoidal method using measurements until 4 hours following the meal. The standardized AUC is the total AUC divided by elapsed time. Those parameters were analyzed analogous to the primary endpoint using an ANCOVA model with treatment group as a factor, and corresponding Baseline postprandial profile as a continuous covariate. This analysis used observed values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 52
Population: MM Population: all participant who participated in the MM tolerance test substudy and who had valid baseline assessments and Week 52 assessments for at least 1 of the MM lab parameters of insulin, proinsulin. The MM tolerance test was performed only in those participants who additionally consented to participate in.
Measure: Least Squares Mean (Standard Error); unit: picomoles/Liter (pmol/L)
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 8 | 16 | 20
picomoles/Liter (pmol/L)
  4hr Ins AUC | 49.2 (50.12) | 2.9 (36.44) | 39.9 (32.62)
  4hr Pro-Ins AUC | 1.0 (17.57) | 1.9 (13.25) | -10.7 (11.62)

13. Secondary Outcome: Albiglutide Plasma Concentration at Weeks 8 and 24
Description: Albiglutide plasma concentration data was analyzed at Week 8 pre-dose, Week 8 post dose, Week 24 pre-dose and Week 24 post-dose. All participants who received albiglutide were initiated on a 30mg weekly dosing regimen; however, beginning at Week 12, participants in the albiglutide 50 mg treatment group were uptitrated to receive albiglutide 50 mg for the remainder of the study.
Time Frame: Weeks 8 and 24
Population: ITT population. Only those participants with a PK sample available for analysis at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Albiglutide 30 mg | Albiglutide 50 mg
Number analyzed (Participants) | 87 | 85
nanograms/milliliter (ng/mL)
  Week 8 Pre-dose, n=85, 85 | 1582 (735) | 1433 (736)
  Week 8 Post-dose, n=87, 80 | 1900 (1093) | 1759 (861)
  Week 24 Pre-dose, n=79, 74 | 1912 (966) | 3060 (1610)
  Week 24 Post-dose, n=81, 72 | 2289 (1255) | 3484 (2301)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs, defined as those events that had a start date on or after the first day of study medication and within 56 days after the end of study medication (up to Week 156), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Albiglutide 30 mg | Albiglutide 50 mg
Serious Adverse Events (participants affected / at risk) | 16/101 | 15/101 | 14/99
Other Adverse Events (participants affected / at risk) | 78/101 | 84/101 | 83/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | Albiglutide 30 mg (N=101) | Albiglutide 50 mg (N=99)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Ischemic stroke (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Drowning (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | Albiglutide 30 mg (N=101) | Albiglutide 50 mg (N=99)
Upper Respiratory tract infection (Infections and infestations) | 17 | 11 | 17
Bronchitis (Infections and infestations) | 10 | 8 | 7
Nasopharyngitis (Infections and infestations) | 6 | 8 | 7
Influenza (Infections and infestations) | 3 | 8 | 6
Cellulitis (Infections and infestations) | 2 | 8 | 2
Sinusitis (Infections and infestations) | 8 | 6 | 7
Urinary tract Infection (Infections and infestations) | 8 | 5 | 7
Gastroenteritis viral (Infections and infestations) | 1 | 4 | 1
Pharyngitis (Infections and infestations) | 7 | 3 | 4
Tinea pedis (Infections and infestations) | 1 | 3 | 1
Ear infection (Infections and infestations) | 3 | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 2 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 2
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Labyrinthitis (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 10 | 14 | 11
Diarrhoea (Gastrointestinal disorders) | 15 | 13 | 16
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 6 | 5 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 4
Constipation (Gastrointestinal disorders) | 4 | 3 | 6
Haemorrhoids (Gastrointestinal disorders) | 4 | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 11 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 6 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Injection site reaction (General disorders) | 2 | 10 | 18
Fatigue (General disorders) | 5 | 7 | 5
Oedema peripheral (General disorders) | 3 | 6 | 4
Injection site rash (General disorders) | 0 | 5 | 3
Injection site erythema (General disorders) | 1 | 4 | 3
Chest pain (General disorders) | 2 | 3 | 1
Injection site haematoma (General disorders) | 5 | 2 | 2
Injection site pruritus (General disorders) | 2 | 2 | 3
Asthenia (General disorders) | 2 | 1 | 2
Irritability (General disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 19 | 15 | 11
Dizziness (Nervous system disorders) | 7 | 5 | 2
Paraesthesia (Nervous system disorders) | 1 | 3 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 2
Sensory Loss (Nervous system disorders) | 3 | 1 | 0
Migraine (Nervous system disorders) | 3 | 0 | 2
Diabetic neuropathy (Nervous system disorders) | 3 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 6 | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 3 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Gout (Metabolism and nutrition disorders) | 1 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 12 | 11 | 12
Hot Flush (Vascular disorders) | 0 | 3 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 4 | 4 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 4 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 1 | 3
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 5 | 4 | 5
Anxiety (Psychiatric disorders) | 1 | 2 | 3
Diabetic retinopathy (Eye disorders) | 1 | 4 | 1
Cataract (Eye disorders) | 2 | 2 | 3
Vision blurred (Eye disorders) | 0 | 1 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 2
Glycosylated haemoglobin increased (Investigations) | 3 | 1 | 0
Angina pectoris (Cardiac disorders) | 5 | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3
Hepatic steatosis (Hepatobiliary disorders) | 3 | 1 | 1
Seasonal allergy (Immune system disorders) | 3 | 1 | 1
Haematuria (Renal and urinary disorders) | 4 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.